CLINICAL TRIAL: NCT04757168
Title: Changes in Regional and Global Cardiac Contractility After Stimulation in Scar Zone with the NOGA System
Acronym: SCARPACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0513
Record Dates: First submitted 2021-02-04; First posted 2021-02-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction
Keywords: stimulation in cardiac scar area
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NOGA TM probe (Experimental)
  Interventions: Device: NOGA TM probe

INTERVENTIONS:
Device: NOGA TM probe — Each subject will be his own witness since the linear local shortening (LLS) will be measured successively in all patients before, then after stimulation of the scar zone (comparison of LLS measured in sinus rhythm then during stimulation in the scar zone for each patient.
  Each subject being his own witness and the two recordings being made a few minutes apart, during the same procedure.

SUMMARY:
Despite a decrease in voltage amplitude in post-infarction scar areas, greater voltage amplitudes are sometimes observed at the time of local extrasystoles mechanically induced by catheters.

However, no study has investigated whether these electrical changes are associated with mechanical changes in local contractility.

However, the voltage is closely correlated to the local contractile function as evidenced by the use of the NOGA system.

ELIGIBILITY:
Inclusion Criteria:

- Patients who should undergo ventricular tachycardia (VT) ablation after a myocardial infarction according to current recommendations, namely: patients with ischemic heart disease (ICD) and with episodes of sustained ventricular tachycardia responsible for internal electric shocks by the implantable automatic defibrillator (ICD) (grade IB recommendation)

OR

* patients with an MIC and an ICD, presenting a first episode of sustained ventricular tachycardia (grade IIa, B recommendation)
* Affiliated with a social protection scheme
* Having signed an informed consent

Exclusion Criteria:

* Contraindication or non-indication for ventricular tachycardia ablation
* Women who are pregnant or of childbearing age and without contraception, breastfeeding women
* Patients without ischemic heart disease
* Patients under guardianship, curatorship or legal protection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of LLS (linear local shortening) via the NOGATM system in percentage | 1month
  Study the change in percentage of LLS during stimulation in a post-infarction scar zone identified by voltage mapping of the left ventricle with the NOGA system, compared to LLS in the same zone measured in atrial stimulation

SECONDARY OUTCOMES:
Evolution of global systolic function: left ventricular ejection fraction | 1month
  Compare the left ventricular ejection fraction (in percentage) during stimulation in a scar area compared to a normal rhythm
Evolution of the global systolic function: integral time velocity under aortic Translation results Evolution of the global systolic function: integral time velocity under aortic | 1month
  Compare the integral time velocity under aortic (in centimeter) during stimulation in a scar area compared to a normal rhythm
Evolution of the global systolic function: strain longitudinal global | 1month
  Compare the strain longitudinal global(in percentage) during stimulation in a scar area compared to a normal rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Anne ROLLIN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- ROLLIN Anne, Toulouse, CHU de Toulouse, France

IPD SHARING:
Plan to Share IPD: No